CLINICAL TRIAL: NCT02119026
Title: A Phase II Study to Assess Efficacy and Safety of Capecitabine and Irinotecan Plus Bevacizumab Followed by Capecitabine and Oxaliplatin Plus Bevacizumab or the Reverse Sequence in Patients With Metastatic Colorectal Cancer
Brief Title: Efficacy And Safety Of Xeliri + Avastin Followed By Xelox + Avastin Or Reverse Sequence In Metastatic Colorectal Cancer
Acronym: PASSION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Werner Scheithauer (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Werner Scheithauer, Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML25153_PASSION
Record Dates: First submitted 2014-04-01; First posted 2014-04-21 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; Patients with metastatic colorectal cancer who did not receive; systemic treatment for their metastatic disease
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: XELIRI + BEV Followed by XELOX + BEV (Active Comparator): capecitabine and irinotecan (XELIRI) plus bevacizumab (AVASTIN; BEV)
  Capecitabine : 800mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on day 1 q3w combined with irinotecan 200mg/m2 iv. d 1 q3w . Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression irinotecan will be replaced by oxaliplatin (arm A). Bevacizumab will be continued.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Irinotecan
- B: XELOX + BEV followed by XELIRI + BEV (Active Comparator): capecitabine and oxaliplatin (XELOX) plus bevacizumab (Avastin; BEV)
  Arm B:
  Capecitabine: 1000mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on d1 q3w combined with oxaliplatin 130mg/m2 iv. d 1 q3w Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression oxaliplatin will be replaced by irinotecan (arm B). Bevacizumab will be continued.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — 800mg/m2 bid d1-14
  ± 1000 mg/m2 bid,days 1-14 q3w: maintenance
  Other Names: Brand Name: Xeloda
  Arms: A: XELIRI + BEV Followed by XELOX + BEV
Drug: Capecitabine — 1000mg/m2 bid d1-14,
  Other Names: Brand name: Xeloda
  Arms: B: XELOX + BEV followed by XELIRI + BEV
Drug: Bevacizumab — 7,5 mg/kg given on d1 q3w
  Other Names: Brand name: Avastin
Drug: Oxaliplatin — 130mg/m2 iv. d 1 q3w
  Arms: B: XELOX + BEV followed by XELIRI + BEV
Drug: Irinotecan — 200mg/m2 iv. d 1 q3w .
  Arms: A: XELIRI + BEV Followed by XELOX + BEV

SUMMARY:
Since its introduction, 5-fluorouracil (5-FU) has been the cornerstone of treatment for metastatic colorectal cancer (mCRC). Meanwhile the oral 5FU pro-drug Capecitabine (Xeloda®) proved equivalence to 5-FU and is a well tolerated alternative combination partner for Irinotecan (XELIRI) or Oxaliplatin (XELOX) which are widely used for first line treatment of mCRC. Recent advances in molecular biology have resulted in the development of an inhibitor of the vascular endothelial growth factor (VEGF) by the monoclonal humanized antibody bevacizumab (Avastin®).

XELOX or XELIRI +bevacizumab have been investigated in several trials, but not in an approach with clearly defined cross-wise XELIRI-XELOX change criteria. This trial investigates two different sequential treatment options with XELIRI/ XELOX in first and second line with the addition of bevacizumab and tries to give answer to the question if there is an optimal sequence for the benefit of the patient.

This is a prospective, randomized, open-label, 2-arm pilot trial in patients with mCRC who did not receive systemic treatment for their metastatic disease. The study is designed to evaluate the efficacy of XELIRI followed by XELOX and XELOX followed by XELIRI + bevacizumab in terms of Duration of Disease Control (DDC).

Patients will be treated with an established first line therapy consisting of either XELOX or XELIRI + bevacizumab. The chemotherapy treatment will be given for 6 months except prior disease progression, unacceptable toxicity or patient refusal. Bevacizumab will be given until disease progression, unacceptable toxicity or patient refusal.

Capecitabine can be given in addition at the investigators' discretion until disease progression, unacceptable toxicity or patient refusal.

If serious side effects occur despite adequate dose reduction, Oxaliplatin or Irinotecan should be discontinued. In case of Oxaliplatin or Irinotecan-related discontinuation Capecitabine and Bevacizumab should be continued. If Capecitabine also has to be discontinued in first line treatment bevacizumab should be continued. In case of permanent discontinuation of bevacizumab for toxicities, chemotherapy should be continued.

Upon completion of first line chemotherapy patients with disease control will receive bevacizumab maintenance treatment. On investigators decision patients can receive Capecitabine as additional maintenance treatment.

The primary endpoint is to determine the efficacy of a modified XELIRI + bevacizumab followed by XELOX + bevacizumab scheme at progression in comparison with the reverse sequence based on DDC.

Secondary endpoints are first line progression-free survival (PFS), second line PFS, overall response rate, time to response, duration of response, overall survival, tumor assessments (based on RECIST criteria) using CT scans, MRI scans, X-ray, bone scan, clinical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age >=18 years
3. Patient must be able to comply with the protocol
4. Histologically or cytologically confirmed carcinoma of the colon and/or rectum with evidence of metastases. 5 )Diagnosis of metastatic disease according to Response Evaluation Criteria in Solid Tumours (RECIST) not more than 3 months prior to enrolment.

6) Life Expectancy of at least 3 months 7) At least one measurable metastatic lesion (as per RECIST criteria) 8) Prior adjuvant or neo-adjuvant chemotherapy/radiotherapy allowed if completed more than 6 months before inclusion. 9) Eastern Collaborative Oncology Group (ECOG) performance score of 0 or 1 10) Adequate haematological function: absolute neutrophil count (ANC) >= 1.5 x 109/L; platelets >= 100 x 109/L, Hb >= 9 g/dL 11) international normalized ratio (INR) <=1.5 and activated partial thromboplastin time (aPTT) <=1.5 x ULN within 7 days prior to starting study treatment 12) Adequate liver function: Serum bilirubin <=1.5 x ULN; alkaline phosphatase and transaminases <=2.5 x ULN (in case of liver metastases < 5 x ULN) 13) Serum Creatinine <=1.5 x ULN 14) Urine dipstick for proteinuria < 2+. If urine dipstick is >= 2+, 24- hour urine must demonstrate <=1 g of protein in 24 hours 15) Negative serum pregnancy test within 7 days of starting study treatment in pre- menopausal women and women < 2 years after the onset of menopause. This test has to be reconfirmed by a urine test, should the 7 days window be exceeded. Fertile women (<2 years after last menstruation) and men must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile).

Exclusion Criteria:

1. Prior chemotherapeutic treatment for metastatic CRC
2. Symptomatic central nervous system (CNS) metastases
3. Significant vascular disease (e.g. aortic aneurysm potentially requiring surgical intervention, pulmonary embolism or recent peripheral arterial thrombosis) within 6 months prior start of study treatment.
4. History of haemoptysis (= a half teaspoon of bright red blood per episode) within 1 month prior start of study treatment
5. Past or current history (within the last 2 years prior to treatment start) of other malignancies (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
6. Clinically significant cardiovascular disease, for example central venous access (CVA) (<=6 months before treatment start), myocardial infarction (<=6 months before treatment start), unstable angina, New York Heart Association (NYHA) >= grade 2, congestive heart failure (CHF), arrhythmia requiring medication, or uncontrolled hypertension.
7. Prior history of hypertensive crisis or hypertensive encephalopathy
8. Treatment with any other investigational agent or any other biological agent (e.g.cetuximab), or participation in another clinical trial within 30 days prior to entering this study.
9. Known hypersensitivity to any of the study drugs
10. Current or recent (within 10 days of first dose of study treatment) chronic use of aspirin (> 325 mg/day)
11. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic (as opposed to prophylactic) purposes.
12. Evidence of bleeding diathesis or coagulopathy.
13. Serious, non healing wound, ulcer, or bone fracture.
14. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment, or anticipation of the need for major surgery during the course of the study. If central venous access device (CVAD) is required for chemotherapy administration, it should be inserted within 2 days prior to study treatment cycle.
15. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior start of study therapy
16. History of abdominal fistula, trachea-oesophageal fistula or any grade 4 non gastrointestinal fistula, gastrointestinal perforation or intra-abdominal abscess before 1st line therapy.
17. History or evidence upon physical/neurological examination of CNS disease (unrelated to cancer) (unless adequately treated with standard medical therapy) e.g. uncontrolled seizures
18. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications
19. Patients with contraindication for cross over chemotherapy (e.g. patients treated with irinotecan based first line therapy and serious polyneuropathy > grade 1, not feasible for oxaliplatin based cross over second line therapy, or patients treated with oxaliplatin based first line therapy and hereditary fructose intolerance not feasible for Irinotecan based cross over second line therapy)
20. Pregnancy or lactation
21. Fertile women (<2 years after last menstruation) and men not willing to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Scheithauer, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Arnold D, Petersen , Kindler M, et al. Patterns of maintenance treatment (Tx) following firstline bevacizumab (bev) plus chemotherapy (CT) for metastatic colorectal cancer (mCRC): Results from a large German community-based cohort study. J Clin Oncol 29: 2011 (suppl 4; abstr 502)
- [Background] Benbow U, Maitra R, Hamilton JW, Brinckerhoff CE. Selective modulation of collagenase 1 gene expression by the chemotherapeutic agent doxorubicin. Clin Cancer Res. 1999 Jan;5(1):203-8. PMID 9918220
- [Background] Yalcin S, Uslu R, Dane F, et al. A Randomized, multicenter phase III trial of bevacizumab plus capecitabine were given as maintenance treatment after initial treatment with bevacizumab plus XELOX in previously untreated metastatic colorectal cancer. J Clin Oncol 29: 2011 (suppl 4; abstr 474)
- [Background] Warren RS, Yuan H, Matli MR, Gillett NA, Ferrara N. Regulation by vascular endothelial growth factor of human colon cancer tumorigenesis in a mouse model of experimental liver metastasis. J Clin Invest. 1995 Apr;95(4):1789-97. doi: 10.1172/JCI117857. PMID 7535799
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] The Criteria Committee of the New York Heart Association. Diseases of the Heart and Blood Vessels: Nomenclature and Criteria for Diagnosis. 6th ed. Boston, MA: Little Brown, 1964
- [Background] Tabernero J, Aranda E, Gomez A, et al. Phase III study of first-line XELOX plus bevacizumab (BEV) for 6 cycles followed by XELOX plus BEV or single-agent (s/a) BEV as maintenance therapy in patients (pts) with metastatic colorectal cancer (mCRC): The MACRO Trial (Spanish Cooperative Group for the Treatment of Digestive Tumors [TTD]). Clin Oncol 28:7s, 2010 (suppl; abstr 3501), Abstract No: 3501
- [Background] Souglakos J, Androulakis N, Syrigos K, Polyzos A, Ziras N, Athanasiadis A, Kakolyris S, Tsousis S, Kouroussis Ch, Vamvakas L, Kalykaki A, Samonis G, Mavroudis D, Georgoulias V. FOLFOXIRI (folinic acid, 5-fluorouracil, oxaliplatin and irinotecan) vs FOLFIRI (folinic acid, 5-fluorouracil and irinotecan) as first-line treatment in metastatic colorectal cancer (MCC): a multicentre randomised phase III trial from the Hellenic Oncology Research Group (HORG). Br J Cancer. 2006 Mar 27;94(6):798-805. doi: 10.1038/sj.bjc.6603011. PMID 16508637
- [Background] Simmonds PC. Palliative chemotherapy for advanced colorectal cancer: systematic review and meta-analysis. Colorectal Cancer Collaborative Group. BMJ. 2000 Sep 2;321(7260):531-5. doi: 10.1136/bmj.321.7260.531. PMID 10968812
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] A. C. Reinacher-Schick, S. Kubicka, W. Freier, et al. Activity of the combination of bevacizumab (Bev) with capecitabine/irinotecan (CapIri/Bev) or capecitabine/oxaliplatin (CapOx/Bev) in advanced colorectal cancer (ACRC): A randomized phase II study of the AIO Colorectal Study Group (AIO trial 0604). J Clin Oncol 26: 2008 (May 20 suppl; abstr 4030)
- [Background] Mabro M, Artru P, Andre T, Flesch M, Maindrault-Goebel F, Landi B, Lledo G, Plantade A, Louvet C, de Gramont A. A phase II study of FOLFIRI-3 (double infusion of irinotecan combined with LV5FU) after FOLFOX in advanced colorectal cancer patients. Br J Cancer. 2006 May 8;94(9):1287-92. doi: 10.1038/sj.bjc.6603095. PMID 16622455
- [Background] Koopman M, Antonini NF, Douma J, Wals J, Honkoop AH, Erdkamp FL, de Jong RS, Rodenburg CJ, Vreugdenhil G, Loosveld OJ, van Bochove A, Sinnige HA, Creemers GM, Tesselaar ME, Slee PHTJ, Werter MJ, Mol L, Dalesio O, Punt CJ. Sequential versus combination chemotherapy with capecitabine, irinotecan, and oxaliplatin in advanced colorectal cancer (CAIRO): a phase III randomised controlled trial. Lancet. 2007 Jul 14;370(9582):135-142. doi: 10.1016/S0140-6736(07)61086-1. PMID 17630036
- [Background] Kim KJ, Li B, Winer J, Armanini M, Gillett N, Phillips HS, Ferrara N. Inhibition of vascular endothelial growth factor-induced angiogenesis suppresses tumour growth in vivo. Nature. 1993 Apr 29;362(6423):841-4. doi: 10.1038/362841a0. PMID 7683111
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Hedrick E, Kozloff M, Hainsworth J, et al. Safety of bevacizumab plus chemotherapy as firstline treatment of patients with metastatic colorectal cancer: Updated results from a large observational registry in the US (BRiTE). J Clin Oncol 2006;24:Abstract 3536.
- [Background] Grothey A, Sargent D, Goldberg RM, Schmoll HJ. Survival of patients with advanced colorectal cancer improves with the availability of fluorouracil-leucovorin, irinotecan, and oxaliplatin in the course of treatment. J Clin Oncol. 2004 Apr 1;22(7):1209-14. doi: 10.1200/JCO.2004.11.037. PMID 15051767
- [Background] Gerber HP, Ferrara N. Pharmacology and pharmacodynamics of bevacizumab as monotherapy or in combination with cytotoxic therapy in preclinical studies. Cancer Res. 2005 Feb 1;65(3):671-80. PMID 15705858
- See also: ethical review committee — http://ethikkommission.meduniwien.ac.at/
- See also: Regulatory authority Austria — http://www.basg.gv.at
- See also: Medical University Vienna/Clin. Division of Oncology — http://www.meduniwien.ac.at/innere-med-1/onkologie/

RESULTS

PARTICIPANT FLOW:
Groups:
- A: XELIRI + BEV Followed by XELOX + BEV: capecitabine and irinotecan (XELIRI) plus bevacizumab (AVASTIN; BEV))
  Capecitabine : 800mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on day 1 q3w combined with irinotecan 200mg/m2 iv. d 1 q3w . Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression irinotecan will be replaced by oxaliplatin (arm A). Bevacizumab will be continued.
  Capecitabine: 800mg/m2 bid d1-14
  ± 1000 mg/m2 bid,days 1-14 q3w: maintenance
  Bevacizumab: 7,5 mg/kg given on d1 q3w
  Irinotecan: 200mg/m2 iv. d 1 q3w .
- B: XELOX + BEV Followed by XELIRI + BEV: capecitabine and oxaliplatin (XELOX) plus bevacizumab (Avastin; BEV))
  Arm B:
  Capecitabine: 1000mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on d1 q3w combined with oxaliplatin 130mg/m2 iv. d 1 q3w Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression oxaliplatin will be replaced by irinotecan (arm B). Bevacizumab will be continued.
  Capecitabine: 1000mg/m2 bid d1-14,
  Bevacizumab: 7,5 mg/kg given on d1 q3w
  Oxaliplatin: 130mg/m2 iv. d 1 q3w
Period: 1st-line Treatment
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Started | 58 | 62
Completed | 32 | 24
Not Completed | 26 | 38
Not completed — Adverse Event | 9 | 14
Not completed — Physician Decision | 3 | 8
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Patient condition or compliance | 6 | 4
Not completed — Surgery of metastases | 2 | 1
Not completed — Death | 2 | 1
Period: 2nd-line Treatment
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Started | 32 | 24
Completed | 23 | 22
Not Completed | 9 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- A: XELIRI + BEV Followed by XELOX + BEV: capecitabine and irinotecan (XELIRI) plus bevacizumab (AVASTIN; BEV)
  Capecitabine : 800mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on day 1 q3w combined with irinotecan 200mg/m2 iv. d 1 q3w . Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression irinotecan will be replaced by oxaliplatin (arm A). Bevacizumab will be continued.
  Capecitabine: 800mg/m2 bid d1-14
  ± 1000 mg/m2 bid,days 1-14 q3w: maintenance
  Bevacizumab: 7,5 mg/kg given on d1 q3w
  Irinotecan: 200mg/m2 iv. d 1 q3w .
- B: XELOX + BEV Followed by XELIRI + BEV: capecitabine and oxaliplatin (XELOX) plus bevacizumab (Avastin; BEV)
  Arm B:
  Capecitabine: 1000mg/m2 bid d1-14, bevacizumab 7,5 mg/kg given on d1 q3w combined with oxaliplatin 130mg/m2 iv. d 1 q3w Bevacizumab (7.5 mg/kg q3w) ± Capecitabine (1000 mg/m2 bid, days 1-14 q3w) maintenance
  At disease progression oxaliplatin will be replaced by irinotecan (arm B). Bevacizumab will be continued.
  Capecitabine: 1000mg/m2 bid d1-14,
  Bevacizumab: 7,5 mg/kg given on d1 q3w
  Oxaliplatin: 130mg/m2 iv. d 1 q3w
- Total: Total of all reporting groups
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV | Total
Number analyzed (Participants) | 58 | 62 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.03 (9.82) | 64.06 (9.70) | 64.53 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 39 | 43 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 58 | 62 | 120

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Duration of Disease Control by Tumor Assessment (CT/MRI/Clinical Examination)
Description: The primary variable was duration of disease control (DDC) and was defined as the sum of progression free survival intervals during first line and second line treatment (= time from the beginning of first line treatment until onset of progression during second line treatment). Patients without progression at the last tumor assessment date during their study participation were censored at this last tumor assessment date (exception: availability of validated information about a later onset of progression or a longer progression free interval - in such a case the date of the follow-up assessment was either defined as the onset of progression or replaced the last tumor assessment date).
Time Frame: screening, every 8 to 9 weeks until progression, at end of treatment (other than progression), every 3 months until progression, death or up to 24 months (whatever comes first)
Population: ITT-Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 58 | 62
days | 373.00 [321.52 to 424.48] | 370.00 [253.255 to 486.745]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.967, Mantel Haenszel

2. Secondary Outcome: First Line Progression Free Survival (PFS)
Description: The first line PFS was defined as the progression free survival interval during first line treatment. Patients without progression at the last tumor assessment date during their study participation were censored at this last tumor assessment date (exception: availability of validated information about a later onset of progression or a longer progression free interval - in such a case the date of the follow-up assessment was either defined as the onset of progression or replaced the last tumor assessment date). Missing onset of progression data because of refusal or because of death was replaced. If several response evaluations for a patient showed progressive disease (PD), the time to PD was assessed by using the first of these measurements.
Time Frame: at progression of disease (PD) in first line therapy or at 28 days safety follow-up in cases without PD
Population: ITT-Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 58 | 62
days | 241 [203.841 to 278.159] | 280 [233.398 to 326.602]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.474, Mantel Haenszel

3. Secondary Outcome: Second Line PFS
Description: The second line PFS was defined as the progression free survival interval during second line treatment. Patients without progression at the last tumor assessment date during their study participation were censored at this last tumor assessment date (exception: availability of validated information about a later onset of progression or a longer progression free interval - in such a case the date of the follow-up assessment was either defined as the onset of progression or replaced the last tumor assessment date). Missing onset of progression data because of refusal or because of death was replaced.
  If several response evaluations for a patient showed progressive disease (PD), the time to PD was assessed by using the first of these measurements.
Time Frame: at progression of disease (PD) in second line therapy or at 28 days safety follow-up in cases without PD
Population: ITT-Population after cross-over
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 32 | 24
days | 129 [60.34 to 197.660] | 155 [108.19 to 201.81]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.464, Mantel Haenszel

4. Secondary Outcome: Overall Response Rate (Number of Participants With Response)
Description: The rate of overall response was measured as the response rate from randomization until the day of documented complete response (CR) or partial response (PR) (whichever status is recorded first).
Time Frame: at the day of documented complete or partial response or at 28 days safety follow-up in cases without PD
Population: ITT-Population
Measure: Count of Participants; unit: Participants
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 58 | 62
Participants | 32 | 36
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.854, Fisher Exact

5. Secondary Outcome: Time to Response
Description: Time to overall response was measured from the time of randomization until the day of documented complete response (CR) or partial response (PR) (whichever status is recorded first). Patients without response were censored at the date of the last tumor assessment, the date of death or the date of refusal.
Time Frame: at the day of documented complete or partial response or at 28 days safety follow-up in cases without PD
Population: ITT-Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 58 | 62
days | 185.0 [97.423 to 272.577] | 178.0 [127.949 to 228.051]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.728, Mantel Haenszel

6. Secondary Outcome: Duration of Response
Description: Duration of overall response was measured from the time that measurement criteria are met for complete response (CR) or partial response (PR) (whichever status was recorded first) until the onset of progression. Patients without progression at the last tumor assessment date during their study participation were censored at this last tumor assessment date (exception: availability of validated information about a later onset of progression or a longer progression free interval - in such a case the date of the follow-up assessment was either defined as the onset of progression or replaced the last tumor assessment date).
  Missing onset of progression data because of refusal or because of death was replaced.
  If several response evaluations for a patient showed progressive disease (PD), the time to PD was assessed by using the first of these measurements.
Time Frame: at the day of documented complete or partial response or at 28 days safety follow-up in cases without PD
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 32 | 36
days | 244.0 [166.888 to 321.112] | 315 [142.297 to 487.703]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.668, Mantel Haenszel

7. Secondary Outcome: Overall Survival of XELIRI Plus Bevacizumab and XELOX Plus Bevacizumab
Description: Overall survival was measured as the time from the randomization date to the date of death. Patients without death date were censored at the date of the last tumor assessment (exception: availability of validated information about a later exitus date or a prolonged survival - in such a case the date of the follow-up assessment was either defined as the exitus date or replaced the last tumor assessment date) or the date of refusal.
Time Frame: date of death or date of last tumor assessment (28d safety f-u) in patients without death
Population: ITT-Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 58 | 62
days | 593.0 [506.691 to 679.309] | 643 [437.227 to 848.773]
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.618, Mantel Haenszel

8. Secondary Outcome: Tumour Assessments (Based on RECIST Criteria) in 1st-line
Description: Best response in first line was based on the tumor assessments (based on RECIST criteria) for target lesions and assessed by CT scans, MRI scans, X-ray, bone scan and clinical examination: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (sum LD) of target lesions; Progressive Disease (PD), >= 20% increase in the sum of the LD of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline, every 8-9 weeks, 28d Safety follow-up
Measure: Number; unit: participants
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 53 | 54
participants
  Progressive Disease (PD) | 4 | 1
  Stable Disease (SD) | 21 | 23
  Partial Response (PR) | 26 | 30
  Complete Response (CR) | 2 | 0
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.792, Wilcoxon (Mann-Whitney) — The rate of overall response was measured as the response rate from randomization until the day of documented complete response (CR) or partial response (PR) (whichever status is recorded first). Analysis corresponds to numbers of CR and PR

9. Secondary Outcome: Tumour Assessments (Based on RECIST Criteria) in 2nd-line
Description: Best response in second line was based on the tumor assessments (based on RECIST criteria) for target lesions and assessed by CT scans, MRI scans, X-ray, bone scan and clinical examination: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (sum LD) of target lesions; Progressive Disease (PD), >= 20% increase in the sum of the LD of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline, every 8-9 weeks, 28d Safety follow-up
Measure: Number; unit: participants
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
Number analyzed (Participants) | 32 | 24
participants
  Progressive Disease (PD) | 7 | 8
  Stable Disease (SD) | 11 | 13
  Partial Response (PR) | 6 | 2
  Complete Response (CR) | 0 | 0
  Not available (NA) | 8 | 1
Statistical Analysis 1: Comparison: A: XELIRI + BEV Followed by XELOX + BEV vs B: XELOX + BEV Followed by XELIRI + BEV; Test type: Superiority; p = 0.371, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: From enrollment until 28 days of last study treatment for the individual patient. Adverse events/serious adverse events still ongoing after that timepoint were followed until last patient last visit (31-Aug-2017).
Description: Clarification regarding threshold for reporting non-serious adverse events: if more than 5 % of patients within on reporting group were affected, non-serious adverse event was reported (more than 3 patients within Arm A and/or Arm B).
Arm/Group | A: XELIRI + BEV Followed by XELOX + BEV | B: XELOX + BEV Followed by XELIRI + BEV
All-Cause Mortality (participants affected / at risk) | 4/58 | 8/62
Serious Adverse Events (participants affected / at risk) | 43/58 | 51/62
Other Adverse Events (participants affected / at risk) | 55/58 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: XELIRI + BEV Followed by XELOX + BEV (N=58) | B: XELOX + BEV Followed by XELIRI + BEV (N=62)
Circulatory collaps (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatectomy (Surgical and medical procedures) | 6 (6) | 8 (9)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Proctectomy (Surgical and medical procedures) | 2 (2) | 2 (2)
Proctocolectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary resection (Surgical and medical procedures) | 2 (2) | 1 (1)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 1 (1)
Sigmoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Thermal ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastates to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 5 (5)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Ulcer (General disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Pain attack (Psychiatric disorders) | 1 (2) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
General physical condition (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal atresia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (8)
Aneamia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 1 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (7)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (4) | 1 (1)
Incarcerated inginual hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Small intestine gangrene (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: XELIRI + BEV Followed by XELOX + BEV (N=58) | B: XELOX + BEV Followed by XELIRI + BEV (N=62)
Hypertension (Vascular disorders) | 13 (23) | 14 (19)
Fatigue (General disorders) | 21 (43) | 27 (63)
General physical health deterioration (General disorders) | 4 (6) | 3 (3)
Mucosal inflammation (General disorders) | 7 (9) | 6 (9)
Oedema (General disorders) | 1 (1) | 4 (8)
Pain (General disorders) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 3 (5) | 5 (9)
Depression (Psychiatric disorders) | 3 (3) | 4 (11)
Insomnia (Psychiatric disorders) | 5 (7) | 3 (3)
Blood pressure increased (Investigations) | 3 (4) | 3 (5)
Body temperature increased (Investigations) | 1 (1) | 4 (4)
C-reactive protein increased (Investigations) | 4 (5) | 10 (15)
Weight decreased (Investigations) | 7 (7) | 14 (19)
Anaemia (Blood and lymphatic system disorders) | 8 (14) | 7 (18)
Neutropenia (Blood and lymphatic system disorders) | 9 (22) | 5 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (15) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Dysgeusia (Nervous system disorders) | 6 (8) | 7 (9)
Headache (Nervous system disorders) | 7 (8) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 6 (7) | 4 (4)
Paraesthesia (Nervous system disorders) | 5 (9) | 7 (10)
Polyneuropathy (Nervous system disorders) | 21 (32) | 37 (90)
Vertigo (Ear and labyrinth disorders) | 8 (9) | 11 (16)
Abdominal pain (Gastrointestinal disorders) | 15 (21) | 11 (15)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 5 (10)
Constipation (Gastrointestinal disorders) | 16 (27) | 14 (18)
Diarrhoea (Gastrointestinal disorders) | 32 (64) | 24 (59)
Flatulence (Gastrointestinal disorders) | 2 (2) | 7 (8)
Nausea (Gastrointestinal disorders) | 21 (38) | 13 (37)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 4 (7)
Vomiting (Gastrointestinal disorders) | 5 (6) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (25) | 5 (5)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (11)
Palmar-plantar erythrodysaestesia syndrome (Skin and subcutaneous tissue disorders) | 20 (46) | 22 (53)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 15 (26) | 11 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 12 (20)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 0 (0)
Nasypharyngitis (Infections and infestations) | 5 (6) | 8 (10)
Rhinitis (Infections and infestations) | 3 (3) | 4 (7)
Urinary tract infection (Infections and infestations) | 11 (13) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT02119026/Prot_SAP_000.pdf